CLINICAL TRIAL: NCT07083349
Title: An Open, Single-Center Exploratory Clinical Study of NK510 Cell Therapy for Refractory Systemic Lupus Erythematosus
Brief Title: NK510 Cell Therapy for Refractory Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Base Therapeutics (Shanghai) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK510-14
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Refractory Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: NK510 is an allogeneic genetically modified NK cell infusion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NK510 infusion (Experimental): NK510
  Interventions: Drug: NK510 : allogeneic genetic modified NK

INTERVENTIONS:
Drug: NK510 : allogeneic genetic modified NK — NK510 is an allogeneic genetic modification of NK cell. NK510 will be administered at a dose of 4x10^7 NK/kg, 8x10^7 NK/kg and 1.2x10^8 NK/kg by a dose-escalation design and administered IV.

SUMMARY:
This is an investigator-initiated, open-label, single-arm study to determine safety and preliminary efficacy of NK510 for the treatment of patients with refractory systemic lupus erythematosus (SLE) in China.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old, male or female.
* A diagnosis of SLE according to the 2019 EULAR (European League Against Rheumatism)/ACR (American College of Rheumatology).
* The subject voluntarily participates in this clinical study and signs the Informed Consent Form (ICF).
* Before screening, the subject must have received glucocorticoid combined with immunosuppressants and/or biological agents for at least 2 months, with a stable dose for more than 2 weeks, but the disease remains active; within 7 days before lymphodepleting conditioning, the blood routine test must meet the following requirements: absolute neutrophil count (ANC) ≥ 1.5×10⁹/L; hemoglobin (Hb) ≥ 80g/L; platelet count (PLT) ≥ 50×10⁹/L.
* SLEDAI-2K score > 8 points at screening.
* Antinuclear antibody (ANA) ≥ 1:80 at screening.
* Having appropriate organ functions:

  1. Liver function: aspartate transaminase (AST) ≤ 3 times the upper limit of normal (ULN); alanine transaminase (ALT) ≤ 3 times ULN; total bilirubin ≤ 1.5 times ULN, unless the subject has a record of Gilbert syndrome; subjects with Gilbert-Meulengracht syndrome with total bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN can be included;
  2. Renal function: serum creatinine ≤ 1.5 times ULN, or creatinine clearance rate ≥ 60 mL/min;
  3. Blood routine: absolute neutrophil count (ANC) ≥ 1.5×10⁹/L; absolute lymphocyte count (ALC) ≥ 0.1×10⁹/L; hemoglobin (Hb) ≥ 80 g/L; platelet count (PLT) ≥ 50×10⁹/L.
* Women of childbearing age must be non-lactating and have a negative serum pregnancy test within 1 week before administration. In addition, all subjects (whether male or female) must agree to use contraception during the period of NK510 treatment starting from enrollment and within 3 months after the end of treatment.
* Able to comply with the study protocol and follow-up procedures.

Exclusion Criteria:

* Patients with active lupus nephritis.
* Those with allergies to the study drug or other medications used in the study protocol.
* Those with any of the following conditions: ① Having received autologous/allogeneic hematopoietic stem cell transplantation within 3 months; ② Having received ultraviolet irradiation therapy within 6 weeks; ③ Having received biologic agent therapy (excluding other medications used in the study protocol) within 4 weeks or 3 half-lives (whichever is longer); ④ Having undergone major surgery or received live vaccines within 4 weeks; ⑤ Having received experimental treatment (except for definite placebo control groups) within 4 weeks.
* Those with other active, known, or suspected autoimmune diseases.
* Presence of uncontrolled active bacterial, viral, fungal, mycobacterial, or other infections requiring treatment with intravenous antibiotics, antiviral drugs, or antifungal drugs within 14 days before lymphodepleting conditioning; however, prophylactic use of these drugs (including intravenous administration) is allowed.
* History of immunodeficiency, including positive HIV test results, or other acquired/congenital immunodeficiency diseases, or history of organ transplantation.
* History of severe cardiovascular and cerebrovascular diseases, including but not limited to: severe cardiac rhythm or conduction abnormalities (e.g., ventricular arrhythmias requiring clinical intervention, third-degree atrioventricular block, etc.); QTc interval > 480 ms on 12-lead electrocardiogram at rest; acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events within 6 months before administration; New York Heart Association (NYHA) cardiac function class ≥ II or left ventricular ejection fraction (LVEF) < 50%.
* Failure to fully recover from major surgery or trauma within 2 weeks before administration.
* History of malignant tumors.
* Screening results of hepatitis B or C virological tests meeting any of the following:

  1. HBsAg positive, and peripheral blood HBV-DNA titer ≥ 1×10³ copies/mL or upper limit of normal;
  2. Anti-HCV positive.
* Those deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Response rate for SLE response index 4 (SRI4) | 3 months, 6 months after the first administration of NK510
  SRI4 response defined as a reduction of ≥4 points on SLEDAI-2000, no new domain A scores and no more than 1 new domain B score on BILAG 2004, and no deterioration in PGA (<0.3 point increase).
Incidence of treatment-related adverse events | 1 year
  This is to measure safety and tolerability of NK510
Dose-limiting toxicity (DLT) rate | 28 days after initial study treatment.
  This is to measure the dose-limiting toxicity of NK510

SECONDARY OUTCOMES:
Number of subjects who achieved lupus low disease activity state (LLDAS) | 3 months, 6 months after the first administration of NK510
  Low lupus disease activity was defined as SLEDAI-2K ≤ 4 points; no major organ system activity, no active hemolytic anemia or gastrointestinal involvement, and no new disease activity manifestations compared with the previous disease assessment; PGA score ≤ 1 point, daily prednisone equivalent dose ≤ 7.5 mg/day, with the permission of using maintenance doses of antimalarials and immunosuppressants (including biological agents).
Number of participants who achieved clinical remission of SLE | 3 months, 6 months after the first administration of NK510
  Clinical remission of SLE was defined by DORIS SLE remission criteria.
The change of SLEDAI-2000(Systemic lupus erythematosus disease activity index 2000) scores | Day 28, 3 months, 6 months after the first administration of NK510
  The change of SLEDAI-2000 score (from 0 to 105 points) will be compared to baseline.
Changes of autoantibody of SLE from baseline | Day 14, 3 months, 6 months after the first administration of NK510
  Autoantibody include anti-dsDNA, anti-nuclear antibody, ANA, anti-Sm antibody, and complement C3, C4.